CLINICAL TRIAL: NCT05845437
Title: A Study on Adequacy of Referrals to Oral and Maxillofacial Surgery Departments in Southern Sweden - Are All Referrals Necessary
Brief Title: On Adequacy of Referrals to Oral and Maxillofacial Surgery
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-01379-01
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Clinical Decision Making; Tooth Extraction; Referral and Consultation; Surgery, Oral; Oral Surgical Procedures
Keywords: Surgery; Dental; Referrals; Relevance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, an ongoing generational shift of the dental community in Sweden originates from an increased number of retiring dentists. Meanwhile, a declining number of dental professionals puts a strain on the care system and reduces the availability of dental care to patients in need of treatment. With fewer experienced dentists, available to guide newly graduated dentists, an increased number of referrals to specialist care units might be a consequence. E.g. referrals to oral and maxillofacial departments originating from a need of assistance in more advanced cases of assessments, treatment planning and therapies. The decreasing number of dentists is also possible to negatively affect the recruitment to specialized dental units, which in turn further decreases treatment availability. When the need for dental care exceeds the capacity of the dental care providers, a possible solution might be to minimize the number of referrals possible to treat in general dentistry, thus prioritize patients truly in need of specialist care. Hence, a reduced waiting time and improved accessibility to an adequate treatment.

The aim of this study is to explore the suitability of referrals concerning exodontia to the departments of oral and maxillofacial surgery in southern Sweden. The primary objective is to assess the level of difficulty in referrals on dental extractions. Secondary objectives are assessments of outcome from treatment and comparison of the suggested treatment of the referral with the outcome. The hypothesis is that the level of difficulty of the required treatments in referrals to oral and maxillofacial departments in southern Sweden is low and constitutes a contributing factor to prolonged waiting queues in specialized dentistry.

DETAILED DESCRIPTION:
The following study is a retrospective study wherein referral letters sent over the course of the months of January to December in 2021 to oral and maxillofacial surgery departments in Lund, Helsingborg and Kristianstad, Sweden will be consecutively collected and reviewed. After a a total screening of referrals concerning dentoalveolar surgery referrals that are related to or possibly related to exodontia will be included into the study. Each referral letter is going to be assessed by the following criteria:

* Patient chief complaint
* Patient's general health
* Tooth/teeth in question
* Clinical assessment
* Radiological assessment
* Diagnosis
* Reason for referral
* Requested treatment: extraction (open or closed), apical surgery, hemisection, consultation, unspecified

The data from referral letters will be compared with data in equivalent journal records of the treatment outcome in every referred case. Each journal record is going to be assessed by the following criteria:

* Patient chief complaint
* Patient's general health
* Tooth/teeth in question
* Clinical assessment
* Radiological assessment
* Diagnosis
* Treatment indication
* Outcome of referral;
* Treatment: extraction (open or closed), apical surgery, hemisection
* No treatment

The level of difficulty of each referred case is going to be measured by a comparison of the referral letters to equivalent patient journal and assessment of treatment outcome. The studied cases will be ranked into one of four categories, wherein categories 1-3 are considered as complicated.

1. Patients whose general heath increases the risk of postoperative medical complications.
2. Cases wherein exodontia cannot be carried out without elevating a surgical flap.
3. Cases wherein exodontia can affect nearby anatomical structures (such as risk of sinus perforation and damage to the inferior alveolar nerve).
4. Otherwise healthy patients where exodontia can be carried out by closed extraction without flap elevation.

Study rational

The recorded data will be analyzed for the level of difficulty, suitability to referral by a comparison with the judged level of difficulty and for the outcome from treatment. Comparisons will be made between the judged level of difficulty with the outcome and the suggested treatment of the referral with the outcome.

Statistical analysis

The sample constitutes of a total inclusion from a cohort limited in time, department and treatment method. The project is designed as an observational trial without control group. Thus, a power-analysis is not valued as necessary for this project.

Simple statistical analysis including mean, standard deviation and range will be used. The limit for statistical significance will be set to p<0.05. A two-sided p-value will be used. Statistical analysis of the data will be performed by use of SPSS - IBM Inc.

Ethical considerations

The study is to be performed in accordance with the 21 CFR, part 50 and the directives laid down in the declaration of Helsinki (Appendix 1 of the declaration, as adopted by the 18th World Medical Assembly, Tokyo, 1975, the 35th WMA, Venice 1983, and the 41st WM A, Hong, Kong 1989, the 48th WMA, Somerset West 1996, the 52nd WMA, Edinburgh 2000 and the clarifications 2002 and 2004).

The project has been submitted to a properly constituted independent Ethics Committee (EC), in agreement with national rules, for formal approval of the study conduct. The decision of the EC concerning the conduct of the study will be in writing to the Investigator and a copy of this decision is archived in the Investigator's Study File.

Patient data protection

The researcher will keep a patient identification list including sufficient information to link records, i.e. CRFs and hospital records. Swedish and local regulations for the handling of computerized data will be followed and described in the written patient information and identification of individual patient data will only be possible for the researcher. A list of the decoded social security numbers of the patients will be kept at the department of Oral and Maxillofacial Surgery, only accessible by the principal researcher.

Report and communication of results After completion of the study, the statistical analysis will be performed by the research group. These data will form the basis for a manuscript intended for publication in a medical journal within two years of the after the project is finished.

Significance and implementation

Adequate referrals are important to have the relatively more expensive specialist health-care units to work as effective as possible. Through a focus of having the best competence predesignated for the most advanced and difficult treatments, the availability and treatment cost will be kept at a desirable level. This is true from both a patient, a health-care provider and a society perspective.

The present study will evaluate the accuracy of the actual referrals in a 12-month time-span. The outcome will give guidance to decision makers in healthcare strategies. Hence, the outcome will, in the short coming future affect education of clinicians, specialist unit geographic establishment and governmental financial support to an improved suitability of health care resources.

The current project aims to clarify the benefits of directed adequate referrals to specialized units of Oral and Maxillofacial Surgery. By knowledge of how the level of existing referrals corresponds to the outcome and how they present, the health care optimization of specialized availability and referral directions will be supported. After publication of the results from the present study, the knowledge will be provided to key decision makers within health care systems.

ELIGIBILITY:
Inclusion Criteria:

- Patients referred for dentoalveolar surgery during 2021.

Exclusion Criteria:

* Word of mouth refferals.
* Referrals send by patients.
* Referrals concerning lesions of the jaw and mucosa that are not of dental origin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Total referred population
Sampling Method: Non-Probability Sample
Enrollment: 624 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Referral question | 12 months
  What is expected from the surgical unit?

SECONDARY OUTCOMES:
Performed treatment | 12 months
  What surgical treatment was given?
Relevance | 12 months
  Was the treatment possible to perform at general dentistry?
Relevance | 12 months
  Was there a discrepancy between expected treatment and performed treatment?

OTHER OUTCOMES:
Content of the referral | 12 Months
  Did the content of the referral meet the need for information?

CONTACTS AND LOCATIONS:
Locations (1):
- Department of oral and maxillofacial surgery, Lund, Skåne County, Sweden